CLINICAL TRIAL: NCT01273545
Title: PRILIGY Usage Patterns in Selected Populations
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Cegedim Strategic Data (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017668; R096769PRE4005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-12-08; First posted 2011-01-10 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Dapoxetine hydrochloride (PRILIGY); Premature ejaculation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Premature Ejaculation | interventions — dapoxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: PRILIGY (dapoxetine hydrochloride) The study will observe characteristics of the patients to whom PRILIGY 30-mg and 60-mg tablets are prescribed in Germany by general practitioners and (separately) by urologists and in Italy by urologists
  Interventions: Drug: PRILIGY (dapoxetine hydrochloride)

INTERVENTIONS:
Drug: PRILIGY (dapoxetine hydrochloride) — The study will observe characteristics of the patients to whom PRILIGY 30-mg and 60-mg tablets are prescribed in Germany by general practitioners and (separately) by urologists, and in Italy by urologists

SUMMARY:
This study will use electronic health services databases to describe the usage patterns of dapoxetine hydrochloride (PRILIGY) in Germany and Italy with a focus on describing the extent and proportion of patients with characteristics suggestive of the use of PRILIGY within, versus outside of the intended use population.

DETAILED DESCRIPTION:
This study will use anonymized (nameless) patient data from electronic health services databases in Germany and Italy to describe the proportion of PRILIGY (dapoxetine hydrochloride) usage among those patients with characteristics suggestive of the use of PRILIGY within versus outside (eg, those with contraindications) of the intended use (IU) population. This is an observational study; no investigational drug will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Received a prescription for PRILIGY
* Treated by physicians who contributed data to the IMS Disease Analyzer database for Germany and Thales database for Italy

Exclusion Criteria:

* Age not specified
* Sex not specified as "male
* " Fewer than 6 months (183 days) of history in the electronic health services databases before receiving the first prescription for PRILIGY (At least 6 months of history in the database is not required for the patients of the German urologists).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male patients prescribed PRILIGY by physicians who contributed data to the CSD electronic health services databases for German urologists, German general practitioners, or Italian general practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-01; Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The proportion patients receiving PRILIGY prescriptions who are within (versus outside of) the IU population. | For up to 1 year

SECONDARY OUTCOMES:
The number of patients prescribed PRILIGY who have conditions or use medications that are described in the special warnings and precautions section of the PRILIGY Summary of Product Characteristics (SPC) | For up to 1 year
The number of patients prescribed PRILIGY who are at risk for bleeding due to current use of nonsteroidal anti-inflammatory drugs (NSAID's) and warfarin. | For up to 1 year
The number of patients prescribed PRILIGY who do not have a diagnosis suggestive of the approved indication. | For up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC C. Clinical Trial, Study Director — Janssen Research & Development, LLC